CLINICAL TRIAL: NCT07257315
Title: Effectiveness of a Program to Improve Balance, Mobility, and Fall Prevention in Older Adults: A Randomized Clinical Trial.
Brief Title: Effectiveness of a Program to Improve Balance, Mobility, and Fall Prevention in Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanidad de Castilla y León (Other)
Responsible Party: Principal Investigator, Jose Angel Delgado Gil, Physical therapist, Sanidad de Castilla y León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2395
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; Risk Factors; Postural Balance; Muscle Strength; Resistance Training Gait; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups. The experimental group performs the Otago Exercise Program in supervised group sessions led by a physiotherapist, while the control group performs the same program independently at home. Each participant remains in their assigned group for the entire duration of the intervention.
Who Masked: Investigator
Masking Description: Outcome assessors are blinded to group assignment. Participants and intervention supervisors are aware of the assigned intervention, but the evaluators measuring functional outcomes, including the Timed Up and Go test and gait speed, do not know which group participants belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Group Otago Exercise Program (Experimental): Participants perform the Otago Exercise Program in supervised group sessions led by a physiotherapist. The program includes structured strength, balance, and functional exercises designed to reduce fall risk. Sessions are conducted 2-3 times per week, and participants follow the program under professional guidance throughout the intervention period.
  Interventions: Behavioral: Otago Exercise Program - Supervised Group
- Home-Based Otago Exercise Program (Active Comparator): Participants perform the same Otago Exercise Program independently at home, following standard written instructions. The program includes the same strength, balance, and functional exercises, performed 2-3 times per week, without direct supervision from a physiotherapist.
  Interventions: Behavioral: Otago Exercise Program - Home-Based

INTERVENTIONS:
Behavioral: Otago Exercise Program - Supervised Group — Participants perform the Otago Exercise Program in supervised group sessions led by a physiotherapist. The program includes structured strength, balance, and functional exercises conducted 2-3 times per week throughout the intervention period.
  Arms: Supervised Group Otago Exercise Program
Behavioral: Otago Exercise Program - Home-Based — Participants perform the same Otago Exercise Program independently at home, following standard written instructions. Exercises include strength, balance, and functional components, performed 2-3 times per week without supervision.
  Arms: Home-Based Otago Exercise Program

SUMMARY:
This trial evaluates the effectiveness of the Otago Exercise Program in adults aged 65 and older. It compares supervised group-based training with an unsupervised home-based version of the same program. The primary aim is to assess changes in Timed Up and Go performance and gait speed before and after the intervention.

DETAILED DESCRIPTION:
This study investigates the effectiveness of the Otago Exercise Program (OEP) as a fall-prevention intervention in adults aged 65 years and older. The OEP is a structured, evidence-based program that includes strength, balance, and functional training exercises designed to reduce fall risk in older adults.

Participants will be randomly assigned to one of two groups. The experimental group will complete the Otago program in supervised group sessions led by a physiotherapist. The control group will perform the same Otago exercises individually at home without supervision, following standard instructions for independent implementation.

The primary objective of the study is to compare the effect of the supervised group-based program versus the unsupervised home-based program on functional mobility and gait performance. Primary outcomes include changes in the Timed Up and Go (TUG) test and gait speed measured before and after the intervention period.

This trial aims to determine whether supervised group training provides additional benefits over independent home-based execution of the Otago program in improving mobility and reducing fall risk among community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older.
* Community-dwelling individuals able to ambulate independently (with or without assistive devices).
* Ability to understand instructions and follow the exercise program.
* Able to attend assessment sessions at baseline and post-intervention.

Exclusion Criteria:

* Severe cognitive impairment that limits ability to follow instructions.
* Medical conditions contraindicating exercise (e.g., unstable cardiac disease, uncontrolled hypertension).
* Recent lower-limb fracture or surgery within the last 6 months.
* Neurological conditions significantly affecting gait or balance (e.g., advanced Parkinson's disease, recent stroke).
* Participation in another structured exercise or fall-prevention program during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | Baseline and immediately after the intervention period (3 months)
  Functional mobility is assessed using the Timed Up and Go test. Participants rise from a chair, walk 3 meters, turn, walk back, and sit down. The time to complete the task is recorded in seconds.
Gait Speed | Baseline and immediately after the intervention period (3 months)
  Walking speed is measured over a standardized distance (6 meters). The participant walks at a comfortable pace, and the time to complete the distance is recorded to calculate gait speed in meters per second.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Angel Delgado-Gil, PT (Physiotherapist), Principal Investigator — Sanidad de Castilla y León
Locations (1):
- Health centre "La palomera", León, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to share individual participant data.